CLINICAL TRIAL: NCT01404000
Title: Phase II Study Exploring Efficacy and Safety of Iodinated Activated Charcoal in COPD
Brief Title: Treatment of Chronic Obstructive Pulmonary Disease (COPD) With Iodinated Activated Charcoal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaLundensis AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PL0801
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iodinated Active Charcoal (Active Comparator): Iodinated activated charcoal 3 gram daily in the morning for 56 days +- 2 days (=8 weeks)
  Interventions: Drug: Iodinated Active Charcoal (IodoCarb)
- non-iodinated activated charcoal (Placebo Comparator): 3g non-iodinated activated charcoal is given daily for 8 weeks
  Interventions: Drug: Iodinated Active Charcoal (IodoCarb)

INTERVENTIONS:
Drug: Iodinated Active Charcoal (IodoCarb) — 3 g will be given as an oral suspension once daily for 56 days

SUMMARY:
The purpose of this study s to determine whether treatment with Iodinated Active Charcoal can improve lung function and physical capacity in patients with chronic obstructive lung disorders. The rational for the study is the observation that COPD patients have an increased tissue load of mercury interfering with the function by NeuroEpithelial Endocrine (NEE) cells in the respiratory tract. Mercury binding to these NEE cells leads to an increased smooth muscle tonus and a reduced response to bronchodilator treatment. Initial observational data have shown an improved lung function and improved functional capacity after treatment motivating a larger placebo controlled POC study

ELIGIBILITY:
Inclusion Criteria:

* Male and >1 year post-menopausal, or surgically sterile female.
* 45-80 years old.
* Smokers and ex-smokers, at least 15 pack years.
* COPD according to GOLD II. FEV% < 70 Post beta2-agonist FEV1 >50 < 80 % of predicted value
* CO diffusion capacity < 75 %.
* Active symptomatic COPD with a COPD assessment test (CAT) score >10.

Exclusion Criteria:

* Alpha-1 antitrypsin deficiency
* Iodine allergy
* Abnormal thyroid function
* Severely reduced kidney function (Cystatin C > 1.5 mg/L.
* Exacerbation within 4 weeks prior to the study.
* Use of per oral steroids within 4 weeks prior to the study.
* Alcohol/drug abuse.
* Psychiatric disease.
* Severe cardio-vascular or other severe disease, according to the clinical investigator.
* Oxygen treatment.
* Participation in another ongoing clinical trial or participation in drug

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Exercise Endurance time (EET) on constant workload 75% of maximum capacity | At baseline and after 8 weeks intervention
  Bicycle work load where the endurance time is recorded. The patients are first doing a maximal workload test determining peak oxygen uptake.

SECONDARY OUTCOMES:
Change in lung function FEV / FVC | At baseline and after 8 weeks intervention
  Change in FEV and FVC in the morning before and after bronchodilation with SABA.
HrQoL | At baseline and after 8 weeks intervention
  SGRQ CAT
Test of thyroid function | At baseline and after 8 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Leif Bjermer, MD Professor, Principal Investigator — Dept of Respiratory Medicine & Allergology, Skane UNiversity Hospital, Lund, Sweden
Locations (1):
- Dept of Respiratory Medcine & Allergology, Skane University Hospital, Lund, Sweden